CLINICAL TRIAL: NCT05124301
Title: Neural Basis of Sensory and Motor Learning: Functional Connections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Hannah Justine Block, Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13138; R01NS112367-01A1 (NIH)
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Basic Science

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perceptual learning (Experimental): Reaching task in which visual information about target finger position is offset to induce a change in perception of the finger.
  Interventions: Behavioral: Perceptual learning

INTERVENTIONS:
Behavioral: Perceptual learning — Reaching task with visual feedback offset from target finger position.

SUMMARY:
The purpose of this study is to understand how the sensory and motor areas of the brain work together to keep a person's hand movements accurate (sensorimotor learning). The investigators hope this information may be useful one day to improve rehabilitation techniques in patients with brain lesions.

DETAILED DESCRIPTION:
Human perception of hand position is multisensory. The brain can estimate it visually, from an image on the retina, and proprioceptively, from receptors in the joints and muscles. The sensory inputs determining these percepts are subject to changes in environmental factors (e.g., lighting) and internal factors (e.g., movement history). Multisensory integration of visual and proprioceptive estimates gives us flexibility to cope with such changes. For example, washing dishes with the hands immersed in water creates a spatial misalignment between vision and proprioception, as water refracts light. The brain resolves this conflict by realigning visual and/or proprioceptive estimates of hand position, and also by adjusting motor commands (visuomotor adaptation). The neural basis of these adaptive processes is poorly understood. The purpose of this study is to find out if multisensory and visuomotor learning are accompanied by changes in resting state connectivity between sensory regions of the brain and other areas.

The first session is a familiarization session for functional magnetic resonance imaging (fMRI) and the behavioral task, and is expected to last 30-40 minutes. Subjects will first fill out screening forms to confirm the answers given during the initial screening, and the Edinburgh handedness inventory to quantify their handedness. If subjects are still eligible, subjects will lie in a mock scanner and perform the functional task: Subjects will have their left index finger taped to a wooden stick, and an experimenter from the team will manipulate the finger with the stick outside of the scanner. Subjects will respond to the different movements by pressing buttons with their right hand. Subjects will also be introduced to the behavioral task, which is performed at an apparatus in the room next to the scanner: Subjects sit in front of a touchscreen and point to targets seen in a mirror.

If subjects are interested in moving on to the main session at this point, the main session will be scheduled.

The main session will take about 2 hours. Subjects will first fill out the MR safety screening form. Subjects will then perform some practice trials of the behavioral task to remind the subject of the task. This will be followed by the first resting state scan (12 min), a 20-30 minute baseline block of the behavioral task (no learning), a second resting state scan (12 min), the 20-30 minute learning block of the behavioral task, and a third resting state scan (12 min). Finally, the subject will do the functional task in the scanner (same as familiarization session, 12 min. total) and an anatomical scan (~6 minutes). The session will conclude with some questions about the subject's subjective experience of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-45 years old
* Right-handed.
* Free of Covid symptoms in week preceding testing.

Exclusion Criteria:

* metallic, mechanical, or magnetic implants;
* are claustrophobic, or are unable to remain still for long periods of time;
* use an intra-uterine device (IUD) whos MR compatibility has not been established.
* Women who are pregnant or think they might be pregnant will also be excluded, as effects of fMRI on the unborn are not known.
* People who have a BMI over 30 will be excluded as it may be uncomfortable or impossible to lay in the MRI scanner and reach the button box.
* Potential subjects will be excluded if they have any neurological disorders, or orthopedic or pain conditions in the upper limbs.
* Investigators will also exclude subjects who do not have normal vision, or corrected-to-normal vision with contacts, or the imaging center does not have a pair of MRI compatible glasses that fits their prescription.
* investigators will invite subjects to reschedule if they have any of the common Covid symptoms within the last week and if they haven't been fully vaccinated or obtained a negative Covid test within the past 4 days. If they don't believe they can meet these criteria on another date, they will be excluded.
* After giving their consent, participants may be excluded during the study if they are unable to perform the tasks or follow instructions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Block, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results published in peer-reviewed journals will be shared except individual brain scans.
Supporting Information: Analytic Code
Time Frame: The data will become available when group results are published in peer-reviewed journals
Access Criteria: Data will be available on www.osf.io for anyone who wishes to download it. The relevant osf registry will be cited in the peer-reviewed publication so that interested readers can find it.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through flyers posted in the community that invited people to contact the study team.
Period: Overall Study
Arm/Group | Perceptual Learning
Started | 76
Completed | 68
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Perceptual Learning
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 44
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76
Edinburgh handedness inventory [Mean (Standard Deviation); unit: units on a scale] — Questionnaire to assess handedness. The scale ranges from -100 (fully left handed) to 100 (fully right handed).
  units on a scale | 90.6 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Resting-state PMv-M1 Functional Connectivity (Fisher Z-transformed Correlation)
Description: Brain activity was measured during a 12-minute resting-state functional magnetic resonance imaging (fMRI) scan. Resting-state functional connectivity between the ventral premotor cortex (PMv) and primary motor cortex (M1) was quantified as the Pearson correlation coefficient between the mean blood-oxygen-level-dependent (BOLD) time series extracted from anatomically defined PMv and M1 regions of interest. Correlation coefficients were Fisher z-transformed to improve normality. For each participant, connectivity values were averaged across all scans acquired during the main session. The outcome measure is the mean Fisher z-transformed correlation value (unitless). Numbers range from -1 (opposite activity in the two regions) to 1 (similar activity in the two regions), with 0 implying no relationship between the two regions.
Time Frame: 3 scans during the main session (2 hours)
Population: 55 is the number of participants who completed the final version of the study.
Measure: Mean (Standard Deviation); unit: unitless (Fisher z-score)
Arm/Group | Perceptual Learning
Number analyzed (Participants) | 55
unitless (Fisher z-score) | 0.64 (0.13)

2. Primary Outcome: Weighting of Vision vs. Proprioception
Description: Measured by comparing where subjects point on the touchscreen when they are estimating visual vs. proprioceptive targets. A person who relies only on vision would have a weighting value of 100%. A person who relies only on proprioception would have a weighting of 0%. A value of 50% would imply equal reliance on vision and proprioception.
Time Frame: Measured during the main session (2 hours)
Population: 55 is the number of participants who completed the final version of the study.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Perceptual Learning
Number analyzed (Participants) | 55
Percent | 43.9 (23.4)
Statistical Analysis 1: Comparison: Perceptual Learning; Tests whether resting state functional connectivity (outcome variable 1) is related to weighting of vision vs. proprioception (outcome variable 2); Test type: Other; p = 0.0022, Regression, Linear; Slope = 0.11

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during each study visit: the familiarization session (about 1 hour) and the main session (about 2.5 hours).
Arm/Group | Perceptual Learning
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT05124301/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT05124301/ICF_001.pdf